CLINICAL TRIAL: NCT03721484
Title: CINtec PLUS Triage of HPV Positive Women in HPV Primary Screening
Brief Title: CINtec PLUS Triage in HPV Primary Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Health and Social Care Trust (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Dr. Mary McMenamin, Dr., Western Health and Social Care Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: v1.0
Record Dates: First submitted 2018-10-17; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CINtec PLUS — CINtec PLUS testing will be used to triage HPV positive women to colposcopy

SUMMARY:
Prospective study which will recruit participants when they attend for a routine cervical screening. The study will evaluate the use of CINtec PLUS for triage of human papillomavirus (HPV) positive participants in HPV primary screening.

DETAILED DESCRIPTION:
The study will recruit participants (9800) prospectively by verbal invitation from the sample taker when they attend for their cervical screening test. Recruitment will take up to one year to complete. Participants in the study will undergo primary HPV testing. This will be followed by cervical cytology testing as per the normal National Health Service Cervical Screening Programme (NHSCSP) screening invitation pathway. Participants testing HPV negative will have reached their end point and will exit the study. Participants who test HPV positive will be triaged by cytology (the cytology screening result, available through the NHSCSP screen will be used). Participants with moderate or severe dyskaryosis (high-grade disease) will be immediately referred to colposcopy (as per NHSCSP guidelines) without further testing. Participants with borderline or mild dyskaryosis (low-grade findings) will undergo CINtec PLUS Cytology triage simulation; however, regardless of the CINtec PLUS result, all participants will also be referred to colposcopy as per NHSCSP guidelines. Participants with negative cytology will undergo CINtec PLUS Cytology triage and those testing positive (an indication of increased risk of CIN2+ [high-grade disease]) will be referred to colposcopy. Participants with negative cytology who also test CINtec PLUS negative will only be referred to colposcopy if they have tested positive for HPV16 or HPV18 as these 2 genotypes have been shown to confer an elevated risk for CIN2+ compared with the other HPV types. Participants with negative cytology who also test CINtec PLUS negative and have tested positive for non HPV16 and HPV18 types will undergo repeat HPV testing at 12 months as the low risk of CIN2+ associated with these participants does not justify immediate colposcopy referral and is unlikely to be granted ethical approval.

Clinical outcomes based on colposcopy and/or histology and/or cervical cytology will be recorded. All biopsies will have one slide stained with CINtec Histology (p16). The risk of CIN2+ will be evaluated for all participants in the study. Subsequently, clinical performance of CINtec PLUS Cytology will be evaluated.

This work will also include a cost analysis.

ELIGIBILITY:
Inclusion Criteria:

* Consenting women aged 25y-64y attending for cervical screening

Exclusion Criteria:

* Women aged <25y and >64y

Ages: 25 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9800 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Risk of high-grade disease | 3 years
  CIN2+ diagnosed on biopsy obtained at colposcopy.
Risk of low-grade disease | 3 years
  <CIN2 as determined by colposcopy assessment/biopsy or cytology ≤Mild/HPV negative.

CONTACTS AND LOCATIONS:
Locations (1):
- WHSCT, Londonderry, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No